CLINICAL TRIAL: NCT01824342
Title: An Open Label, Single Arm, Extension Study to Evaluate the Long Term Safety of Denosumab for Prolonging Bone Metastasis-Free Survival in Men With Hormone-Refractory Prostate Cancer
Brief Title: Denosumab for Prolonging Bone Metastasis-Free Survival in Men With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080585; 2010-021846-23 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Castrate-resistant Prostate Cancer
MeSH Terms: interventions — Denosumab

ARMS (1):
- Denosumab (Experimental): Participants received denosumab 120 mg subcutaneously every 4 weeks for up to 3 years in this open-label extension study.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Administered by subcutaneous injection
  Other Names: XGEVA®

SUMMARY:
This is a multi-national, multi-center, open-label, single-arm extension study for the prolongation of bone metastasis-free survival in men with hormone-refractory (androgen independent) prostate cancer. Patients currently participating in the phase 3 study 20050147 (NCT00286091) will be offered this study if a positive benefit:risk compared with placebo is determined in the 20050147 study. The primary endpoint of the 20050147 study is bone metastases-free survival determined by the time to first occurrence of bone metastases (either symptomatic or asymptomatic) or death from any cause. Participants will receive open-label denosumab administered once every 4 weeks (Q4W) subcutaneously (SC) until they developed a bone metastasis or for up to 3 years, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently undergoing every 4 weeks scheduled assessments in the phase 3 study 20050147
* Subjects must sign the informed consent before any study specific procedures are performed

Exclusion Criteria:

* Developed sensitivity to mammalian cell derived drug products during the 20050147 study
* Currently receiving any unapproved investigational product other than denosumab
* Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- Czechia (4):
  - Research Site, Hradec Králové
  - Research Site, Pelhřimov
  - Research Site, Prague
  - Research Site, Tábor
- United Kingdom (4):
  - Research Site, Newcastle
  - Research Site, Northwood
  - Research Site, Sheffield
  - Research Site, Sutton

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-arm, open-label extension (OLE) phase of a phase 3, randomized, double-blind study (Study 20050147; NCT00286091) comparing denosumab with placebo on prolonging bone metastasis-free survival in men with hormone-refractory (androgen independent) prostate cancer.
Pre-assignment Details: All participants received denosumab during the OLE phase; in the parent study participants were initially randomized in a blinded manner to receive denosumab at a dose of 120 mg or placebo every 4 weeks.
Groups:
- Placebo/Denosumab: Participants who received placebo in the parent study received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks (Q4W) for up to 3 years.
- Denosumab/Denosumab: Participants who received denosumab in the parent study received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks (Q4W) for up to 3 years.
Period: Overall Study
Arm/Group | Placebo/Denosumab | Denosumab/Denosumab
Started | 11 | 7
Completed | 2 | 2
Not Completed | 9 | 5
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Disease Progression | 1 | 1
Not completed — Physician Decision | 5 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Denosumab | Denosumab/Denosumab | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (4.3) | 70.3 (7.4) | 71.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 7 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 11 | 7 | 18
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    Grade 0 | 7 | 5 | 12
    Grade 1 | 4 | 1 | 5
    Grade 2 | 0 | 1 | 1
    Grade 3 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0
Albumin-adjusted calcium [Mean (Standard Deviation); unit: mmol/L] | 2.44 (0.10) | 2.42 (0.04) | 2.43 (0.08)
Creatinine [Mean (Standard Deviation); unit: umol/L] | 88.40 (14.25) | 89.66 (23.63) | 88.89 (17.80)
Phosphorus [Mean (Standard Deviation); unit: mmol/L] | 1.09 (0.22) | 1.01 (0.24) | 1.06 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Deaths
Description: A serious adverse event is defined as an adverse event that meets at least one of the following serious criteria: • fatal, • life threatening, • requires in-patient hospitalization or prolongation of existing hospitalization, • results in persistent or significant disability/incapacity, • congenital anomaly/birth defect, and/or • other significant medical hazard. The adverse event severity grading scale used was the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, according to the following: Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE. The investigator assessed whether each adverse event was possibly related to the investigational product (IP).
Time Frame: From the first dose of open-label denosumab until 4 weeks after the last; maximum time on study was 37 months. Follow-up survival information was collected for up to 3 years after the last dose of blinded investigation product in the 20050147 study.
Population: Safety analysis set, which included participants who had properly documented informed consent for protocol 20080585 and received at least 1 dose of open-label denosumab.
Measure: Number; unit: participants
Arm/Group | Placebo/Denosumab | Denosumab/Denosumab
Number analyzed (Participants) | 11 | 7
participants
  Any adverse event (AE) | 11 | 7
  Serious adverse event | 7 | 4
  Fatal adverse event | 2 | 0
  AE leading to study discontinuation | 2 | 1
  AE leading to IP discontinuation | 4 | 1
  CTCAE Grade 3, 4, or 5 | 6 | 2
  AE related to investigational product (IP) | 2 | 3
  Serious AE related to IP | 0 | 2
  Fatal AE related to IP | 0 | 0
  AE related to IP leading to study discontinuation | 1 | 1
  AE related to IP leading to IP discontinuation | 1 | 1
  AE related to IP and CTCAE Grade 3, 4, or 5 | 0 | 1
  Deaths | 4 | 1
  Deaths on study | 2 | 0
  Deaths during the safety follow-up | 2 | 1

2. Primary Outcome: Percent Change From Baseline in Laboratory Values
Time Frame: Baseline and Week 49
Population: Safety analysis set with available laboratory data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Denosumab | Denosumab/Denosumab
Number analyzed (Participants) | 10 | 6
percent change
  Albumin-adjusted Calcium | -0.9 (2.5) | 1.1 (3.1)
  Alkaline Phosphatase | -23.8 (21.8) | -1.6 (20.5)
  Creatinine | 16.3 (31.5) | 2.4 (5.8)
  Phosphorus | -2.6 (25.2) | 0.0 (10.4)

3. Primary Outcome: Number of Participants With Anti-denosumab Neutralizing Antibody Formation
Time Frame: 3 years
Population: Participants exposed to open-label denosumab with ≥ 1 antibody sample
Measure: Number; unit: participants
Arm/Group | Placebo/Denosumab | Denosumab/Denosumab
Number analyzed (Participants) | 10 | 7
participants | 0 | 0

4. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: A scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work); 2 = Ambulatory and capable of all self care, but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry out any self-care. Totally confined to bed or chair; 5 = Dead.
Time Frame: Baseline and Week 49
Population: Safety analysis set with available data at both time points
Measure: Number; unit: participants
Arm/Group | Placebo/Denosumab | Denosumab/Denosumab
Number analyzed (Participants) | 10 | 6
participants
  4-point increase in PS | 0 | 0
  3-point increase in PS | 0 | 0
  2-point increase in PS | 0 | 0
  1-point increase in PS | 0 | 1
  No change | 10 | 5
  1-point decrease in PS | 0 | 0
  2-point decrease in PS | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Placebo/ Denosumab 120 mg Q4W: Participants who received placebo in the parent study received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks (Q4W) for up to 3 years.
- Denosumab/ Denosumab 120 mg Q4W: Participants who received denosumab in the parent study received open-label denosumab 120 mg by subcutaneous injecton once every 4 weeks (Q4W) for up to 3 years.
Arm/Group | Placebo/ Denosumab 120 mg Q4W | Denosumab/ Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 7/11 | 4/7
Other Adverse Events (participants affected / at risk) | 11/11 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ Denosumab 120 mg Q4W (N=11) | Denosumab/ Denosumab 120 mg Q4W (N=7)
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Urinary sediment present (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ Denosumab 120 mg Q4W (N=11) | Denosumab/ Denosumab 120 mg Q4W (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Catheter site pain (General disorders) | 2 | 0
Device expulsion (General disorders) | 1 | 0
Device leakage (General disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Abscess of salivary gland (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Viral infection (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Radiation injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 2 | 2
Urinary sediment present (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 1
Poor quality sleep (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 3 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 1
Nocturia (Renal and urinary disorders) | 2 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Prostatic pain (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.